CLINICAL TRIAL: NCT04435028
Title: Ketotifen: Novel Use as a Cardioprotective Agent in Breast Cancer Patients Receiving Anthracycline-containing Chemotherapy as Well as the Potential Beneficial Effects of Ketotifen in the Hypothetical Management of COVID-19
Brief Title: Ketotifen: as a Cardioprotective Agent in Breast Cancer Patients Receiving Anthracycline-containing Chemotherapy
Status: Completed | Type: Observational
Sponsor: Horus University (Other)
Responsible Party: Principal Investigator, hosny ahmed elewa, head of pharmacy practice department, Horus University
Other Study IDs: 1890-1-2019
Record Dates: First submitted 2020-06-15; First posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Breast Cancer; Iron Chelation
MeSH Terms: conditions — Breast Neoplasms | interventions — Ketotifen

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- control group: 55 patients received their standard therapy (anthracycline-containing chemotherapy without ketotifen)
  Interventions: Drug: Ketotifen 1 MG
- ketotifen group: Ketotifen Group: 56 patients received anthracycline-containing chemotherapy plus ketotifen as a cardioprotective agent. Ketotifen will be given orally as one tablet (1 mg/tablet) 3 times daily, before and during the chemotherapeutic cycle for 6 cycles of treatment
  Interventions: Drug: Ketotifen 1 MG

INTERVENTIONS:
Drug: Ketotifen 1 MG — Ketotifen is added to patients on anthracycline-containing chemotherapy for 6 months
  Other Names: placebo

SUMMARY:
The objective of our study was to evaluate the expected cardioprotective effects of ketotifen due to its activity as an iron-chelating agent previously uncovered by us in the in vitro chemical test which included in the study, when used in patients receiving anthracyclines for the treatment of breast cancer. The study was a randomized : , prospective controlled trial : , and the patients were identified by coded numbers to maintain privacy. Eligible patients (111) fulfilled the criteria. Control Group: 55 patients received their standard therapy (anthracycline-containing chemotherapy without ketotifen). Ketotifen Group: 56 patients received anthracycline-containing chemotherapy plus ketotifen as a cardioprotective agent. Ketotifen will be given orally as one tablet (1 mg/tablet) 3 times daily, before and during the chemotherapeutic cycle for 6 cycles of treatment. Blood samples were obtained from all patients, and echocardiography two times for each patient at baseline and after 6 months (EF%).

DETAILED DESCRIPTION:
The objective of our study was to evaluate the expected cardioprotective effects of ketotifen due to its activity as an iron-chelating agent previously uncovered by us in the in vitro chemical test which included in the study, when used in patients receiving anthracyclines for the treatment of breast cancer. The study was a randomized : , prospective controlled trial : , and the patients were identified by coded numbers to maintain privacy. Eligible patients (111) fulfilled the criteria. Control Group: 55 patients received their standard therapy (anthracycline-containing chemotherapy without ketotifen). Ketotifen Group: 56 patients received anthracycline-containing chemotherapy plus ketotifen as a cardioprotective agent. Ketotifen will be given orally as one tablet (1 mg/tablet) 3 times daily, before and during the chemotherapeutic cycle for 6 cycles of treatment. Blood samples were obtained from all patients, and echocardiography two times for each patient at baseline and after 6 months (EF%).

The aim is to prove and evaluate the prophylasis effect of ketotifin from cardiotoxicity induced by anthracyclines therapy without decreasing the anti-tumor action of anthracycline.

Because coronaviruses theoretically induce iron overload so, ketotifen has a potential beneficial effect in the management of COVID-19 as well.

ELIGIBILITY:
Inclusion Criteria:

* cancer patients receiving anthracycline chemotherapy in their protocol alone (without any cardioprotective agent),
* aged 30-60, and
* female subjects were included as they were female breast cancer patients, and,
* patients who had an adequate baseline echocardiography.

Exclusion Criteria:

* who had a history of heart failure,
* arrhythmia,
* cardiac catheterizations,
* angina,
* uncontrolled hypertension, and
* uncontrolled diabetes,
* patients with impaired liver function tests,
* patients who previously received anthracycline-containing regimens, and
* any cardiotoxic chemotherapy regimens, previous history of chest wall irradiation.
* Brian metastasis.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — as the study was on breast cancer female patients
Study Population: The study participants were recruited from the Oncology Department, Menoufia University Hospital, Egypt. The study was designed and conducted in compliance with the ethical principles of Good Clinical Practice Guidelines and the Declaration of Helsinki
Sampling Method: Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-08-13 (Actual); Study Completion 2019-08-13 (Actual)

PRIMARY OUTCOMES:
prophylaxis effect of Ketotifen on patient's hearts during the treatment of anthracyclines | 6 months
  the serum levels of LDH, CK-MB, troponin I, TIBC, ferritin, anti-cardiolipin IgG, and, iron were done

CONTACTS AND LOCATIONS:
Locations (1):
- Horus University, Damietta, Damiete Governonate, Egypt